CLINICAL TRIAL: NCT01898663
Title: Safety and Therapeutic Efficacy of DCs Vaccine Combined With Cytokine-induced Killer Cells in Patients With AML: a Phase Ⅰ/Ⅱ Study
Brief Title: DCs Vaccine Combined With Cytokine-induced Killer Cells in Patients With AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-DC/CIK
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: High-risk Soft Tissue Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adenovirus-transfected DC + CIK (Experimental): Adenovirus-transfected autologous DCs + CIK cells
  Interventions: Biological: Adenovirus-transfected DC + CIK

INTERVENTIONS:
Biological: Adenovirus-transfected DC + CIK — Adenovirus-transfected autologous DC vaccine plus CIK cells

SUMMARY:
The aim of this Phase Ⅰ/Ⅱ study is to evaluate the safety and efficacy of dendritic cells (DCs) vaccine combined with cytokine-induced killer (CIK) cells in patients with AML. Experimental recombinant adenovirus-transfected DCs, which engineered to express MUC1 and Survivin are used for DCs-based immunotherapy. Based on the results of our previously performed preclinical study with DCs vaccine combined with CIK cells, the investigators plan to perform the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with the diagnosis of AML
* Age≥18 years at time of consent
* KPS(Karnofsky Performance Scale) ≥70
* Patient's written informed consent
* No steroid therapy within 4 weeks of first DC vaccination
* Stable disease, complete response and partial response(WHO, RECIST)
* Predicted survival≥3 months

Exclusion Criteria:

* Serious dysfunction of vital organs(heart, liver or kidney)
* Received organ transplantation
* Patients with other malignancies or brain metastases
* History of autoimmune diseases
* Pregnant and breast-feeding patient
* Active or chronic infectious diseases
* History of allergy or hypersensitivity to study product excipients
* Currently participating in another clinical trial
* Received chemotherapy, radiotherapy, immune inhibitor (such as corticosteroid) or other immunotherapy (such as vaccine) during prior 4 weeks
* Unfit for participating in this clinical trial in investigators' opinions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS/OS | 1 years after DC/CIK treatment

SECONDARY OUTCOMES:
Number of participants with adverse events | 3 days within DC/CIK treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hu, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of Hematopoietic Stem Cell Transplantation, Beijing, China